CLINICAL TRIAL: NCT02866773
Title: Family Holistic Health Community Promotion, A Community-based Research to Promote Healthy Diet and Physical Activity in Hong Kong Island: A Cluster Randomized Controlled Trial (cRCT)
Brief Title: A Community-based Family Holistic Health Promotion Project in Hong Kong: A Cluster Randomized Controlled Trial (cRCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Island Women Association (Unknown); The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Professor Lam Tai-Hing, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW -1622
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Family; Well-being; Physical Activity; Healthy Diet
Keywords: Family; well-being; Physical activity; Diet
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- PA1:Education sessions, Reminders, Whataps group (Experimental): The intervention includes Physical activity knowledge enhancement session, Physical activity anti-inertia Reminders , Physical activity ambassadors' electronic communication group.
  Interventions: Behavioral: PA2: Education sessions, Reminders; Behavioral: PA3: Education sessions, Whataps group; Behavioral: PA4: Education sessions; Behavioral: HD1: Education sessions, Reminders, Whataps group
- PA2:Education sessions, Reminders (Active Comparator): The intervention includes Physical activity knowledge enhancement session and Physical activity anti-inertia Reminders
  Interventions: Behavioral: PA3: Education sessions, Whataps group; Behavioral: PA4: Education sessions
- PA3:Education sessions, Whataps group (Active Comparator): The intervention includes Physical activity knowledge enhancement session and Physical activity ambassadors' electronic communication group.
  Interventions: Behavioral: PA2: Education sessions, Reminders; Behavioral: PA4: Education sessions
- PA4:Education sessions (Active Comparator): The intervention includes Physical activity knowledge enhancement session only.
  Interventions: Behavioral: HD4: Education sessions
- HD1:Education sessions, Reminders, Whataps group (Experimental): The intervention includes Health diet knowledge enhancement session, Health diet anti-inertia Reminders , Health diet ambassadors' electronic communication group.
  Interventions: Behavioral: PA1: Education sessions, Reminders, Whataps group; Behavioral: HD2: Education sessions, Reminders; Behavioral: HD3:Education sessions, Whataps group; Behavioral: HD4: Education sessions
- HD2:Education sessions, Reminders (Active Comparator): The intervention includes Health diet knowledge enhancement session, Health diet anti-inertia Reminders , and Health diet ambassadors' electronic communication group.
  Interventions: Behavioral: HD3:Education sessions, Whataps group; Behavioral: HD4: Education sessions
- HD3:Education sessions, Whataps group (Active Comparator): The intervention includes Health diet knowledge enhancement session and Health diet ambassadors' electronic communication group.
  Interventions: Behavioral: HD2: Education sessions, Reminders; Behavioral: HD4: Education sessions
- HD4:Education sessions (Active Comparator): The intervention includes Health diet knowledge enhancement session only.
  Interventions: Behavioral: HD4: Education sessions

INTERVENTIONS:
Behavioral: PA1: Education sessions, Reminders, Whataps group — The intervention includes three components:
  * Physical activity knowledge enhancement session: one core session and one booster session on increasing physical activity and reducing sedentary behavior
  * Physical activity Anti-inertia Reminder: souvenirs and electronic healthy messages are sent to participants in this group to promote the awareness of performing regular exercise
  * Physical activity ambassadors' electronic communication group: the community leaders and ambassadors' formed an electronic communication group to share their experience on performing regular physical activity and program implementation.
  Arms: HD1:Education sessions, Reminders, Whataps group
Behavioral: PA2: Education sessions, Reminders — The intervention includes two components:
  * Physical activity knowledge enhancement session: one core session and one booster session on increasing physical activity and reducing sedentary behavior
  * Physical activity Anti-inertia Reminder: souvenirs and electronic healthy messages are sent to participants in this group to promote the awareness of performing regular exercise
  Arms: PA1:Education sessions, Reminders, Whataps group; PA3:Education sessions, Whataps group
Behavioral: PA3: Education sessions, Whataps group — The intervention includes two components:
  * Physical activity knowledge enhancement session: one core session and one booster session on increasing physical activity and reducing sedentary behavior.
  * Physical activity ambassadors' electronic communication group: the community leaders and ambassadors' formed an electronic communication group to share their experience on performing regular physical activity and program implementation.
  Arms: PA1:Education sessions, Reminders, Whataps group; PA2:Education sessions, Reminders
Behavioral: PA4: Education sessions — The intervention includes one component only:
  - Physical activity knowledge enhancement session: one core session and one booster session on increasing physical activity and reducing sedentary behavior
  Arms: PA1:Education sessions, Reminders, Whataps group; PA2:Education sessions, Reminders; PA3:Education sessions, Whataps group
Behavioral: HD1: Education sessions, Reminders, Whataps group — The intervention includes two components:
  - Healthy diet knowledge enhancement session: one core session and one booster session on increasing reducing sugary intake.
  Healthy diet Anti-inertia Reminder: souvenirs and electronic healthy messages are sent to participants in this group to promote the awareness of reducing sugary intake.
  - Healthy diet ambassadors' electronic communication group: the community leaders and ambassadors' formed an electronic communication group to share their experience on reducing sugary intake and program implementation.
  Arms: PA1:Education sessions, Reminders, Whataps group
Behavioral: HD2: Education sessions, Reminders — The intervention includes two components:
  * Healthy diet knowledge enhancement session: one core session and one booster session on increasing reducing sugary intake.
  * Healthy diet Anti-inertia Reminder: souvenirs and electronic healthy messages are sent to participants in this group to promote the awareness of reducing sugary intake.
  Arms: HD1:Education sessions, Reminders, Whataps group; HD3:Education sessions, Whataps group
Behavioral: HD3:Education sessions, Whataps group — The intervention includes two components:
  * Healthy diet knowledge enhancement session: one core session and one booster session on increasing reducing sugary intake.
  * Healthy diet ambassadors' electronic communication group: the community leaders and ambassadors' formed an electronic communication group to share their experience on reducing sugary intake and program implementation.
  Arms: HD1:Education sessions, Reminders, Whataps group; HD2:Education sessions, Reminders
Behavioral: HD4: Education sessions — The intervention includes one component only:
  - Healthy diet knowledge enhancement session: one core session and one booster session on increasing reducing sugary intake.
  Arms: HD1:Education sessions, Reminders, Whataps group; HD2:Education sessions, Reminders; HD3:Education sessions, Whataps group; HD4:Education sessions; PA4:Education sessions

SUMMARY:
In Hong Kong, nearly 40% of adults were overweight or obese, and about 60% of total registered deaths were due to four major preventable non-communicable diseases. Many residents are lack of attention to personal healthy lifestyle and family holistic health. This project focuses particularly on the promotion of healthy diet and physical activities enhancement in families through the well-established community network of the Hong Kong Island Women Association (HKIWA). This project includes three major components: Train-the-trainer and -ambassador workshop, community-based family interventions, and public education events. It is expected that knowledge and skills of the community leaders and ambassadors are strengthened through the 'Train-the-trainer and -ambassador' (TTTA) workshops. Furthermore, they are expected to help the implementation of community-based family interventions and public education events on the personal and family holistic health of the community participants.

DETAILED DESCRIPTION:
According to World Health Organization (WHO), the prevalence of obesity among all nations has nearly doubled since 1980. High body mass index (BMI) is one of the major risk factors of many non-communicable diseases (NCD) and is the result of unhealthy diet and physical inactivity. In Hong Kong, the Department of Health (DH) found in 2012, through the telephone surveys, that nearly 40% of adults were overweight or obese. About 60% of total registered deaths in Hong Kong were due to four major preventable NCD, which were cancer, heart diseases, stroke and chronic lower respiratory diseases. Therefore, population-based interventions for collective health benefits, especially regarding weight management, are essential in lowering the risk of NCD in the total population.

Given the high proportion of overweight and obese individuals among the local population, achieving modest or even small behavioral changes in diet or activity could potentially lead to significant improvements in public health. Promotion of healthy diets and physical activity is one of the five recommended cost-effective interventions that have been addressed in The Lancet Series. The implementation of policies to promote healthy diets - reducing sugary beverages, in particular - and physical activity due to the likelihood of wide-ranging health gains, including prevention of overweight and cardiovascular disease, on a population level is advocated.

Facing the same challenges of the rest of the world that many residents are lacking of attention on healthy lifestyle, the Hong Kong SAR Government has a burden to improve the well-being of the general public. The Government has recently established a Committee on 'Reduction of Salt and Sugar in Food'. They will steer the direction, formulate and oversee the Action Plans for Salt and Sugar Reduction in Hong Kong. The aim is to reduce the intake of salt and sugar by residents to meet the WHO recommendations. The Centre for Food Safety showed that carbonated drinks and fruit juices were popular in Hong Kong. However, the added sugar does not have any nutritional value but increases the risk of overweight and obesity. Therefore, the promotion of healthy family diet is appropriate for improving a current public health situation in Hong Kong. On the other hand, the Leisure and Cultural Services Department have been jointed with the Department of Health to launch the 'Healthy Exercise for All Campaign' for raising the public's interest in exercising. However, none of the campaigns have addressed the problems and barriers of the sedentary people and their families. The barriers include myths and wrong perceptions, e.g.; exercise has to be difficult, or one has to find much time, spend much money and do lots of high intensive exercise to be beneficial.

This project is aimed to motivate participants to improve start with 'zero-time exercise' and reduce sugary beverages, which can be incorporated into daily life to reduce day-to-day sedentary time and sugar intake together with family members of all ages, that can then act as a trigger for active and healthy lifestyle. Few exercises can be done by the family members together. The investigators shall motivate participants to share what they have learned with their family members and to do 'zero-time exercise' and reduce sugary beverage's intake together. This project includes three major components: Train-the-trainer and -ambassador workshop, community-based family interventions, and public education events. Knowledge and skills of the community leaders and ambassadors will be strengthened through the 'Train-the-trainer and -ambassador' workshop. The trainees will be expected to help the implementation of community-based family interventions and public education events on the personal and family holistic health of the community participants.

Outcome and process evaluations will be used to assess the engagement, implementation and effectiveness of the project. Focus group and in-depth interviews will be conducted to obtain feedback, and opinion of the community leaders, ambassadors and community participants. Quantitative questionnaire assessments will be conducted at different time points to assess the effectiveness of the project on the key components of personal and family holistic health, and family well-being. The assessment time points are before and immediately after the core session, before and after the booster session at one month, three months, six months for community participants. An additional assessment for the community leaders and ambassadors is nine months.

ELIGIBILITY:
Inclusion criteria

1. Train-the-trainers and ambassador programs:

   * Cantonese speaking
   * Intact verbal and hearing abilities for interpersonal communication
   * Reading and writing abilities for questionnaire completion
   * Community leaders and health ambassadors
   * Aged 18 or above
2. Community-based family interventions:

   * Cantonese speaking
   * Intact verbal and hearing abilities for interpersonal communication
   * Reading and writing abilities for questionnaire completion
   * Aged 12 or above
3. Public education events:

   * Reading and writing abilities for questionnaire completion
   * Aged 12 or above

Exclusion criteria

- Participants who fail to meet the inclusion criteria, or are unable to sign the consent form.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in behaviour | baseline and one month
  Assessed by outcome-based questionnaire

SECONDARY OUTCOMES:
Change in behavior | Baseline, 1 month, 3 months, 6 months, and 9 months
  Assessed by outcome-based questionnaire
Change in learning | Baseline, immediately after core session, 1 month, 3 months, 6 months, and 9 months
  Assessed by outcome-based questionnaire
Influence on family members | Baseline, 1 month, 3 months, 6 months, and 9 months
  Assessed by outcome-based questionnaire
Personal physical and psychological health | Baseline, 1 month, 3 months, 6 months, and 9 months
  Assessed by outcome-based questionnaire
Quality of Life | Baseline, 1 month, 3 months, 6 months, and 9 months
  Assessed by a validated questionnaire (SF12)
Family well-being | Baseline, 1 month, 3 months, 6 months, and 9 months
  Assessed by outcome-based questionnaire
Family relationship | Baseline, 1 month, 3 months, 6 months, and 9 months
  Assessed by outcome-based questionnaire
Satisfaction towards the program | immediately after core session, immediately after booster session at 1 month, 6 months, 9 months
  Assessed by outcome-based questionnaire
Response on Anti-inertia Reminder | 1 months, 3 months, 6 months
  Assessed by outcome-based questions
Social network relationship | 6 months and 9 months
  Assessed by outcome-based questions

CONTACTS AND LOCATIONS:
Overall Officials: Tai-hing Lam, MD, Principal Investigator — School of Public Health, The University of Hong Kong; Piana He, MSc, Study Director — Hong Kong Island Women Association
Locations (1):
- Hong Kong Island Women Association, Hong Kong Island, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Artinian NT, Fletcher GF, Mozaffarian D, Kris-Etherton P, Van Horn L, Lichtenstein AH, Kumanyika S, Kraus WE, Fleg JL, Redeker NS, Meininger JC, Banks J, Stuart-Shor EM, Fletcher BJ, Miller TD, Hughes S, Braun LT, Kopin LA, Berra K, Hayman LL, Ewing LJ, Ades PA, Durstine JL, Houston-Miller N, Burke LE; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing. Interventions to promote physical activity and dietary lifestyle changes for cardiovascular risk factor reduction in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 27;122(4):406-41. doi: 10.1161/CIR.0b013e3181e8edf1. Epub 2010 Jul 12. No abstract available. PMID 20625115
- [Background] Mozaffarian D, Afshin A, Benowitz NL, Bittner V, Daniels SR, Franch HA, Jacobs DR Jr, Kraus WE, Kris-Etherton PM, Krummel DA, Popkin BM, Whitsel LP, Zakai NA; American Heart Association Council on Epidemiology and Prevention, Council on Nutrition, Physical Activity and Metabolism, Council on Clinical Cardiology, Council on Cardiovascular Disease in the Young, Council on the Kidney in Cardiovasc. Population approaches to improve diet, physical activity, and smoking habits: a scientific statement from the American Heart Association. Circulation. 2012 Sep 18;126(12):1514-63. doi: 10.1161/CIR.0b013e318260a20b. Epub 2012 Aug 20. PMID 22907934
- [Background] Haines DJ, Davis L, Rancour P, Robinson M, Neel-Wilson T, Wagner S. A pilot intervention to promote walking and wellness and to improve the health of college faculty and staff. J Am Coll Health. 2007 Jan-Feb;55(4):219-25. doi: 10.3200/JACH.55.4.219-225. PMID 17319328
- [Background] Epstein LH, Paluch RA, Wrotniak BH, Daniel TO, Kilanowski C, Wilfley D, Finkelstein E. Cost-effectiveness of family-based group treatment for child and parental obesity. Child Obes. 2014 Apr;10(2):114-21. doi: 10.1089/chi.2013.0123. Epub 2014 Mar 21. PMID 24655212